CLINICAL TRIAL: NCT04432051
Title: The Significance of Lung Ultrasonography in the Follow-up and Treatment of COVID-19 Patients With Respiratory Failure
Brief Title: The Use of Lung Ultrasonography in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Gaziosmanpasa
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2020-08

CONDITIONS: Ultrasonography
Keywords: lung ultrasonography; intensive care unit; position; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: patients will be divided into two groups, those with and without ultrasound.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRUP Control (Placebo Comparator): The daily respiratory system examination of COVID-19 patients who are hospitalized in the intensive care unit is performed and the necessary mechanical ventilation applications are performed by evaluating the arterial blood gas analysis.
  Interventions: Behavioral: mechanical ventilator settings and position
- GRUP Ultrasonography (Active Comparator): The daily respiratory system examination of COVID-19 patients who are hospitalized in the intensive care unit is performed and the necessary mechanical ventilation applications are performed by evaluating the arterial blood gas analysis. However, the lung of the patient will be evaluated by ultrasound and the position to use the lung capacity most appropriately will be given.
  Interventions: Behavioral: mechanical ventilator settings and position

INTERVENTIONS:
Behavioral: mechanical ventilator settings and position — Mechanical ventilation settings and patient position will be re-evaluated

SUMMARY:
In COVID-19 patients hospitalized in the intensive care unit due to respiratory failure, lung ultrasonography will be tried to be given an appropriate position that will effectively use lung capacity and its effect on oxygenation will be investigated.

DETAILED DESCRIPTION:
In this study, the COVID-19 patients hospitalized in the intensive care unit due to respiratory failure will be evaluated. Participants will be divided into two groups as patients undergoing lung ultrasonography (Group Ultrasonography ) and those without lung ultrasonography (Group Control).

While performing lung ultrasonography, each hemithorax will be evaluated using anterior axillary line and posterior axillary line into anterior, lateral and posterior region, and each region will be divided into 6 quadrants, upper and lower. Each hemithorax will be scanned by the investigators, scored in 6 regions using a convex ultrasonography probe with the Lung Ultrasound Score (LUS score).

Participants in both groups will be evaluated by comparing arterial blood gas analyzes before examination (with/without ultrasonography), at the 2nd and 12th hours. Is there any change in arterial blood gas values such as PO2 and PCO2 at 0, 2 and 12 hours so that oxygenation and ventilation between Group Ultrasonograpy and Group Control will be evaluated?

ELIGIBILITY:
Inclusion Criteria:

* Patients have been diagnosed with COVID 19
* Patients in the intensive care unit over the age of 18

Exclusion Criteria:

* Patients not diagnosed with COVID 19
* Patients with cardiac problems
* Patients with renal problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Change in PO2 values | 12 hours
  Effect of positioning on ultrasound guidance on oxygenation assessed by changes between pO2 values.

SECONDARY OUTCOMES:
Change in PCO2 values | 12 hours
  Effect of positioning on ultrasound guidance on ventilation assessed by changes between pCO2 values.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazoosmanpasa Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No